CLINICAL TRIAL: NCT05461183
Title: Assessment of Cumulative Incidence and Factors Associated With Hospital Re-admission and Severe Maternal Morbidity After Delivery Discharge in British Columbia
Brief Title: Postpartum Outcomes in BC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other)
Responsible Party: Principal Investigator, Marianne Vidler, Assistant Professor, University of British Columbia
Other Study IDs: H21-01696
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Morbidity;Perinatal; Pregnancy Complications; Pregnancy Related
Keywords: severe maternal morbidity; postpartum period; hospital readmission
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Readmission/ SMM post-delivery discharge: All women aged 15-49 who were readmitted up to six weeks post-delivery discharge and/or experienced at least one SMM event up to six weeks post-delivery
  Interventions: Other: Retrospective database analysis
- De novo readmission/ SMM post-delivery discharge: All women aged 15-49 who were readmitted up to six weeks post-delivery discharge and/or experienced at least one SMM event post-delivery, excluding those who experienced a SMM in the two months before delivery or during delivery hospitalization
  Interventions: Other: Retrospective database analysis
- No post-delivery discharge readmission/ SMM at any time (CONTROL): All women aged 15-49 who did not experience post-delivery discharge readmission and/or SMM at any time
  Interventions: Other: Retrospective database analysis

INTERVENTIONS:
Other: Retrospective database analysis — This study will review data provided by the BCPDR from April 1, 2008 to March 31, 2021.

SUMMARY:
For every case of maternal death, many more women experience life-threatening complications during pregnancy and childbirth. Yet, severe maternal morbidity (SMM) cases are often overlooked post-delivery. Women have reported that roughly 15% of SMM cases first occurred in the six weeks following delivery. The underlying factors associated with these morbidities are likely different than those occurring antenatally and at the time of delivery. Further research is required to elucidate the exact burden of SMM in the postpartum period in British Columbia (BC).

DETAILED DESCRIPTION:
The ratio of maternal morbidity to maternal mortality is increasing globally (Geller 2018). In high-income countries, the World Health Organization (WHO) recommends routinely surveilling SMM to assess maternal health and quality of care (Geller 2018). To our knowledge, this is the first study conducted among pregnancies in BC aiming to examine the cumulative incidence, timing, and factors associated with postpartum maternal morbidity and hospital readmissions.

This is a retrospective cohort study will use data from the BC Perinatal Data Registry (BCPDR), which contains maternal, fetal and neonatal health information from 99% of all deliveries in BC. The primary outcome assessed will be the cumulative incidence of hospital readmissions and SMM events occurring after delivery discharge within the first six weeks (42 days) of delivery. Secondary outcomes will include SMM-diagnosis, the rate and timing of postpartum SMM and readmissions, and maternal characteristics associated with these events. A multinominal logistic regression model will examine the association between postpartum SMM or readmission and determinants.

ELIGIBILITY:
Inclusion Criteria:

* Delivered in BC from April 1, 2008 to March 31, 2021
* Consented to data collected by the BCPDR

Exclusion Criteria:

• None

Ages: 15 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Those who delivered between April 1, 2008 to March 31, 2021 using data from the BC Perinatal Data Registry (BCPDR).
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2008-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Maternal hospital readmission | Up to six weeks post-delivery discharge
  Cumulative incidence of women who get readmitted into the hospital after being discharged post-delivery
Severe maternal morbidity (SMM) event | Up to six weeks post-delivery discharge
  Cumulative incidence of women who experience least one SMM event, defined as: severe pre-eclampsia, HELLP, eclampsia; severe haemorrhage; maternal ICU admission; surgical complications; hysterectomy; sepsis; embolism, shock, DIC; assisted ventilation; cardiac conditions; acute renal failure; several uterine rupture; cerebrovascular accidents; and other types of maternal morbidity.

SECONDARY OUTCOMES:
SMM type | Up to six weeks postpartum
  Type of SMM event experienced
Rate of hospital readmission and SMM events | Up to six weeks postpartum
  Frequency of women who get readmitted to the hospital after discharge and/or experienced at least one SMM event
Timing of hospital readmission and SMM events | Up to six weeks postpartum
  Specific time frames for women who get readmitted to the hospital after discharge and/or experienced at least one SMM event
Maternal characteristics | Up to six weeks postpartum
  Characteristics associated with hospital readmission and SMM events after delivery discharge, such as age, race, geographic location, fetal outcome, mode of delivery and pre-existing maternal comorbidities (hypertension, diabetes, and mental health conditions).

REFERENCES:
- [Background] Geller SE, Koch AR, Garland CE, MacDonald EJ, Storey F, Lawton B. A global view of severe maternal morbidity: moving beyond maternal mortality. Reprod Health. 2018 Jun 22;15(Suppl 1):98. doi: 10.1186/s12978-018-0527-2. PMID 29945657
- [Background] Dzakpasu S, Deb-Rinker P, Arbour L, Darling EK, Kramer MS, Liu S, Luo W, Murphy PA, Nelson C, Ray JG, Scott H, VandenHof M, Joseph KS. Severe maternal morbidity surveillance: Monitoring pregnant women at high risk for prolonged hospitalisation and death. Paediatr Perinat Epidemiol. 2020 Jul;34(4):427-439. doi: 10.1111/ppe.12574. Epub 2019 Aug 12. PMID 31407359